CLINICAL TRIAL: NCT07318467
Title: Prophylactic Regimen of Intravenous Oxytocin, Intravenous Tranexamic Acid, and Intramuscular Ergot Derivative for Primary Prevention of Postpartum Hemorrhage in Intrapartum Cesarean Section Versus Intravenous Carbetocin Alone
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Abdalla Mousa, Lecturer of Obstetrics and Gynecology, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MS-306-2025
Record Dates: First submitted 2025-12-20; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Post Partum Hemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Group A will receive a combination regimen of intravenous Oxytocin (5-10IU), Tranexamic acid (intravenous bolus 1 gram), and intramuscular ergot derivative (methylergometrine maleate 0.2 mg/ ml).
  The participants will receive intravenous Oxytocin immediately after delivery of the fetus, intravenous Tranexamic acid during the procedure and intramuscular Ergot derivative after delivery of the placenta
  Interventions: Drug: Intravenous Oxytocin, Intravenous Tranexamic Acid, and Intramuscular Ergot Derivative
- Group B (Active Comparator): Group B will receive intravenous Carbetocin (100 mcg) only. The participants will receive intravenous Carbetocin only immediately after delivery of the fetus.
  Interventions: Drug: Intravenous Carbetocin alone

INTERVENTIONS:
Drug: Intravenous Oxytocin, Intravenous Tranexamic Acid, and Intramuscular Ergot Derivative — Group A will receive a combination regimen of intravenous Oxytocin (5-10IU), Tranexamic acid (intravenous bolus 1 gram), and intramuscular ergot derivative (methylergometrine maleate 0.2 mg/ ml).
  The participants will receive intravenous Oxytocin immediately after delivery of the fetus, intravenous Tranexamic acid during the procedure and intramuscular Ergot derivative after delivery of the placenta
  Arms: Group A
Drug: Intravenous Carbetocin alone — Group B will receive intravenous Carbetocin (100 mcg) only. The participants will receive intravenous Carbetocin only immediately after delivery of the fetus.
  Arms: Group B

SUMMARY:
While Carbetocin is effective in reducing PPH, the combination of oxytocin, Tranexamic acid, and Ergot derivatives may offer additional benefits in high-risk populations. We hypothesize that the combination regimen will reduce PPH incidence and severity compared to Carbetocin alone and may be more cost effective

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing C-Sections.
* Women between the ages of 18 and 45 years.
* Singleton pregnancy.
* Gestational age is equal to or more than 36 weeks.
* No known coagulopathy or bleeding disorders.
* No known hypersensitivity or allergy to drugs used in the study.
* Normal obstetric ultrasonography with no fetal abnormalities.

Exclusion Criteria:

* Hemodynamically unstable or immobile patients.
* Multifetal pregnancy.
* Patients who are receiving prophylactic or therapeutic anticoagulation.
* Known comorbidities and contraindications to the use of Ergot derivatives or Carbetocin such as hypertension or cardiovascular disorders.
* Placenta previa and/or Placenta accreta spectrum.
* History of thromboembolism.
* Preeclampsia or eclampsia.
* Any additional measurements needed to control or stop excessive bleeding intraoperatively such as uterine artery ligation or use of sterile gelatin absorbable foam.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Amount of blood loss | during and up to 24 hours after cesarean section